CLINICAL TRIAL: NCT01689779
Title: Effect of High-dose Cholecalciferol Supplementation on Perioperative Vitamin D Status in Colorectal Surgery Patients
Brief Title: High Dose Preoperative Cholecalciferol Supplementation and Perioperative Vitamin D Status
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bio-Tech Pharmacal, Inc. (Industry)
Responsible Party: Principal Investigator, Sadeq A. Quraishi, Assistant Professor of Anaesthesia, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012P001852
Record Dates: First submitted 2012-09-04; First posted 2012-09-21 (Estimated); Results first posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-08

CONDITIONS: Hypovitaminosis D
Keywords: vitamin D; surgery; acute stress
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Active Comparator): A maximum of 40 patients will receive a one-time oral dose of 100,000 IU cholecalciferol 3-7 days before their scheduled elective surgery.
  Interventions: Drug: 100,000 IU cholecalciferol
- Placebo (Placebo Comparator): A maximum of 40 patients will receive a one-time oral sugar pill 3-7 days before their scheduled elective surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 100,000 IU cholecalciferol — active drug
  Other Names: vitamin D3
  Arms: Cholecalciferol
Drug: Placebo — comparator drug
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
A growing body of evidence suggests that robust postoperative immune function is associated with a lower risk of surgical site infections (SSIs). At the same time, vitamin D is increasingly recognized as a key regulator of the innate and adaptive immune systems. The investigators elected to conduct the current study in patients who will undergo colorectal surgery since these patients are historically at higher risk of developing SSIs and therefore would be ideal for future investigations.

DETAILED DESCRIPTION:
While vitamin D insufficiency [25(OH)D <30 ng/mL] is common in the general population, hypovitaminosis D may affect 40-80% of patients in the perioperative setting. Recent evidence also suggests that surgical stress may be associated with a 40% reduction in circulating 25(OH)D levels when compared to preoperative values. Moreover, the derangement in perioperative 25(OH)D levels may be sustained for up to 3 months after surgery. This finding has potential implications regarding modifiable risk factors for surgical site infections (SSIs), which account for nearly 40% of all nosocomial infections. On aggregate, SSIs result in 3.7 million extra hospital days per annum and an added burden of $1.6 billion in annual healthcare costs. A growing body of evidence suggests that robust postoperative immune function is associated with a lower risk of SSIs. At the same time, vitamin D is increasingly recognized as a key regulator of the innate and adaptive immune systems. Yet, optimization of perioperative vitamin D status remains grossly understudied. Although our overarching aim is to study the impact of vitamin D status on SSIs, the focus of the current investigation is to determine whether the administration of a "bolus" oral dose of cholecalciferol (vitamin D3) in the preoperative setting alters vitamin D status in the perioperative setting (compared to a placebo). The investigators elected to conduct the current study in patients who will undergo colorectal surgery since these patients are historically at higher risk of developing SSIs and therefore would be ideal for future investigations.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* 18 years or older;
* Scheduled for elective (non-emergent) colorectal surgery;
* Cleared for anesthesia; and
* Expected to stay overnight following surgery

Exclusion Criteria:

* Scheduled for a purely laparoscopic procedure;
* Diagnosis of a terminal illness and/or in hospice care;
* Inability to sign informed consent;
* Inability to comply with study protocol;
* Intending to start vitamin D supplementation within 30 days of surgery;
* Intending to leave the Boston area during the follow-up period;
* History of renal stones or hypercalcemia;
* Medical conditions that can cause hypercalcemia (e.g. metastatic cancer, sarcoidosis, myeloma primary hyperparathyroidism)
* History of hypercalcemia
* History of severe anemia (Hematocrit <25%)
* Medications that affect vitamin D metabolism (e.g. anti-epileptics, tuberculosis medication); and
* Already enrolled or planning to enroll in a research study that would conflict with full participation in the current study or confound the observation or interpretation of the study findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sadeq A Quraishi, MD, MHA, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cholecalciferol: 40 patients will receive 100,000 IU cholecalciferol orally 3-7 days before surgery.
  100, 000 IU cholecalciferol
- Sugar Pill: 40 patients will receive a sugar pill orally 3-7 days before surgery.
  Placebo: sugar pill
Period: Overall Study
Arm/Group | Cholecalciferol | Sugar Pill
Started | 28 | 32
Completed | 28 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol | Sugar Pill | Total
Number analyzed (Participants) | 28 | 32 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (13) | 61 (13) | 57 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 25 | 28 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent (%) Change in 25(OH)D 5 Days Following Supplementation With 100,000 IU Cholecalciferol
Description: 3-7 days before surgery, patients will receive 100,000 IU of cholecalciferol (vs. placebo) during their pre-op assessment. They will also have their baseline vitamin D status measured during this initial visit. The main study outcome is to determine if 100,000 IU cholecalciferol can be given preoperatively to safely boost vitamin D status. To assess vitamin D status, we will measure: 1) 25(OH)D and 2) LL37
Time Frame: Patients will be followed between the initial preoperative evaluation day and an average duration of 5 days
Population: Data are presented as percent change in levels between baseline assessment and day of surgery
Measure: Mean (Standard Deviation); unit: percent change in 25(OH)D
Arm/Group | Cholecalciferol | Sugar Pill
Number analyzed (Participants) | 28 | 32
percent change in 25(OH)D | 8 (6) | -2 (4)

2. Secondary Outcome: Percent (%) Change in Pre-surgical 25(OH)D Within 24 Hours of Surgery
Description: The goal is to determine whether pre-operative supplementation with 100,000 IU cholecalciferol (vs. placebo) alters the natural course of short-term changes in vitamin D status following surgery. To assess vitamin D status, we will measure: 1) 25(OH)D and 2) LL37.
Time Frame: Patients will be followed between the day of surgery and 1 day after surgery
Population: Data are presented as percent change in levels between baseline assessment and day after surgery
Measure: Mean (Standard Deviation); unit: Percent change in 25(OH)D
Arm/Group | Cholecalciferol | Sugar Pill
Number analyzed (Participants) | 28 | 32
Percent change in 25(OH)D | -5 (6) | -4 (4)

3. Other Pre Specified Outcome: Percent (%) Change in Pre-surgical 25(OH)D 2 Weeks After Surgery
Description: The goal is to determine whether pre-operative supplementation with 100,000 IU cholecalciferol (vs. placebo) alters the natural course of changes in vitamin D status within 10-18 days after surgery. To assess vitamin D status, we will measure: 1) 25(OH)D and 2) LL-37.
Time Frame: Patients will be followed between the day of surgery and an average duration of 14 days after surgery
Population: Data are presented as percent change in levels between baseline assessment and 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: Percent change in 25(OH)D
Arm/Group | Cholecalciferol | Sugar Pill
Number analyzed (Participants) | 28 | 32
Percent change in 25(OH)D | 3 (7) | 1 (11)

4. Primary Outcome: Percent (%) Change in LL-37 5 Days Following Supplementation With 100,000 IU Cholecalciferol
Description: as for outcome 1
Time Frame: Patients will be followed between the initial preoperative evaluation day and an average duration of 5 days
Population: Data are presented as percent change in levels between baseline assessment and day of surgery
Measure: Mean (Standard Deviation); unit: percent change in LL-37
Arm/Group | Cholecalciferol | Sugar Pill
Number analyzed (Participants) | 28 | 32
percent change in LL-37 | -10 (17) | -5 (12)

5. Secondary Outcome: Percent (%) Change in Pre-surgical LL-37 Within 24 Hours of Surgery
Description: as for outcome 2
Time Frame: Patients will be followed between the day of surgery and 1 day after surgery
Population: Data are presented as percent change in levels between baseline assessment and day after surgery
Measure: Mean (Standard Deviation); unit: Percent change in LL-37
Arm/Group | Cholecalciferol | Sugar Pill
Number analyzed (Participants) | 28 | 32
Percent change in LL-37 | -3 (24) | -5 (31)

6. Other Pre Specified Outcome: Percent (%) Change in Pre-surgical LL-37 2 Weeks After Surgery
Description: as for outcome 3
Time Frame: Patients will be followed between the day of surgery and an average duration of 14 days after surgery
Population: Data are presented as percent change in levels between baseline assessment and 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: Percent change in LL-37
Arm/Group | Cholecalciferol | Sugar Pill
Number analyzed (Participants) | 28 | 32
Percent change in LL-37 | 16 (27) | 2 (37)

ADVERSE EVENTS:
Time Frame: Data was collected over a period of 30 days post drug administration
Arm/Group | Cholecalciferol | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 1/28 | 1/32
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/32
Other Adverse Events (participants affected / at risk) | 0/28 | 0/32

LIMITATIONS AND CAVEATS:
A small sample size and a relatively homogenous patient cohort at a major teaching hospital limit the generalizability of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No